CLINICAL TRIAL: NCT01053338
Title: Open Label,Balanced,Randomized,Two-treatment,Two-sequence,Two Period,Single-dose,Crossover Oral Bioequivalence Study of Ibuprofen and Diphenhydramine Citrate 200mg/38mg Caplets of Dr.Reddy's and Advil®PM of Wyeth in Normal,Healthy,Adult,Human Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Dr.Reddy's Ibuprofen and Diphenhydramine Citrate 200 mg/38 mg Caplets Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Director Clinical Pharmacology & Pharmacokinetics, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 155-07
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioequivalence,Ibuprofen Diphenhydramine Citrate,Crossover
MeSH Terms: interventions — Ibuprofen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen and Diphenhydramine Citrate (Experimental): Ibuprofen and Diphenhydramine Citrate 200 mg/38 mg Caplets of Dr. Reddy's
  Interventions: Drug: Ibuprofen and Diphenhydramine Citrate
- Advil (Active Comparator): Advil PM 200 mg/38 mg Tablets of Wyeth
  Interventions: Drug: Ibuprofen and Diphenhydramine Citrate

INTERVENTIONS:
Drug: Ibuprofen and Diphenhydramine Citrate — Ibuprofen and Diphenhydramine Citrate 200mg/38mg Caplets
  Other Names: Advil PM

SUMMARY:
To determine the single-dose oral bioequivalence study of Ibuprofen and Diphenhydramine citrate 200 mg/38 mg caplets of Dr. Reddy's Laboratories Limited, India and Advil®PM, of Wyeth consumer health care, USA, in normal, healthy, adult, human subjects under fed conditions.

DETAILED DESCRIPTION:
Detailed Description : The study was conducted as an Open label, balanced, randomized, two-treatment, two-sequence, two period,single-dose, crossover oral bioequivalence study of Ibuprofen and Diphenhydramine citrate 200 mg/38 mg caplets of Dr. Reddy's Laboratories Limited, India and Advil@PM, of Wyeth Consumer Healthcare, USA., in normal, healthy, adult, human subjects under fed conditions. A total number of forty (40) subjects were enrolled in the study and all the subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects aged between 18 and 45 years (including both).
* Subjects with a BMI between 18.5 - 24.9 Kg/m2 (including both) but body weight not less than 45 Kgs.
* Subjects with normal health as determined by personal medical history, clinical examination, and laboratory examinations including serological tests.
* Subjects having normal 12 lead electrocardiogram (ECG).
* Subjects having normal chest X-Ray (P/A view).
* Subjects able to communicate effectively.
* Subjects willing to give written informed consent and adhere to all the requirements of this protocol.
* Female subjects who are postmenopausal or surgically sterile.
* Female subjects practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm,intrauterine device (IUD) or abstinence.

Exclusion Criteria:

* Subjects having contraindications or hypersensitivity to Ibuprofen Diphenhydramine citrate or related group of drugs.
* History or presence of any medical conditions or disease according to the opinion of the physician.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 10 cigarettes or bidis/day or consumption of tobacco products).
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Systolic blood pressure less than 90 mm Hg or more than 140 mm Hg.
* Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50 beats/minute or more than 100 beats/minute.
* Use of any prescribed medication during last two weeks or OTC medicinal products during the last one week preceding the first dosing.
* Major illness during 3 months before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breast-feeding.
* Female subjects with child bearing potential using prohibited contraceptive method (Oral, Injectable or Implantable hormonal agents).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study of Dr. Reddys Laboratories Limited, Ibuprofen and Diphenhydramine Citrate Caplets under fasting condition | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: N. Netaji, MD, Principal Investigator — GVK Biosciences Pvt. Ltd
Locations (1):
- GVK Biosciences Pvt. Ltd, Amīrpet, Hyderabad, India